CLINICAL TRIAL: NCT00035360
Title: Phase 3 Study of PEG-Intron in Heavily Treatment-experienced, HIV-infected Patients
Brief Title: Phase III PEG-Intron in HIV-infected Patients (Study P00738)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00738
Record Dates: First submitted 2002-05-02; First posted 2002-05-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections; AIDS
Keywords: PEG-Intron; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — peginterferon alfa-2b

INTERVENTIONS:
Drug: PEG-Intron

SUMMARY:
This is a randomized, double-blind, multicenter trial testing 2 doses of PEG-Intron, 1.0mcg/kg/week and 3.0mcg/kg/week in heavily treatment-experienced HIV-infected patients compared to placebo. The study will evaluate the efficacy and safety of PEG-Intron when added to stable optimized background antiretroviral therapy in this patient population.

DETAILED DESCRIPTION:
This study will randomize 675 patients (225 in each of the 3 arms) to either: PEG-Intron 1mcg; 3mcg or Placebo, at 90 centers worldwide. Each center will enroll approximately 10 patients.

Study drug will be added to optimized background anti-retroviral therapy of patients whose HIV RNA is incompletely suppressed by their therapy (HIV RNA 400-50,000 copies/ML) after 2-6 months.

A single dose reduction of 50% will be allowed for toxicity. An Interim Analysis will be conducted when 50% of patients have completed 24 weeks of therapy. The study treatment phase will be 48 weeks with monthly visits for virologic virologic and safety monitoring. The primary endpoint is change in HIV RNA from baseline to week to assess efficacy. Durability of response will be assessed at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* History of virologic failure on at least 2 antiretroviral regimens including exposure to at least one NRTI, one NNRTI and one PI
* HIV RNA >400-<50,000 copies/mL
* Laboratory parameters: platelet count (75,000u/L, hemoglobin >9gm/dl, absolute neutrophil count >1,000/uL, SGOT/SGPT<5xULN.

Exclusion Criteria:

* Current ribavirin therapy
* Subjects with a recent diagnosis or history of moderate or severe depression requiring ongoing psychiatric intervention
* Females of childbearing potential who are breastfeeding, who are pregnant, or not using adequate birth control measures
* Concomitant use of immunosuppressants or cytotoxic agents
* History of seizure disorder requiring use of anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html